CLINICAL TRIAL: NCT05267184
Title: Swedish Trial on Embolization of Middle Meningeal Artery Versus Surgical Evacuation in Chronic Subdural Hematoma
Acronym: SWEMMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Sahlgrenska University Hospital (Other); Karolinska University Hospital (Other); Norrlands University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/02670
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-11

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Trephining

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: telephone interview at 3 and 12 months by clinical outcomes assessor blinded to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization of middle meningeal artery (Experimental): Participants receive endovascular treatment with embolization of the middle meningeal artery ipsilaterally to the chronic subdural hematoma(s).
  Interventions: Procedure: Endovascular treatment of the middle meningeal artery
- Standard neurosurgical hematoma evacuation and drainage (Active Comparator): Participants receive standard neurosurgical hematoma evacuation via burr hole or mini craniotomy and post-operative subdural or subgaleal drainage.
  Interventions: Procedure: Standard neurosurgical hematoma evacuation

INTERVENTIONS:
Procedure: Endovascular treatment of the middle meningeal artery — The middle meningeal artery on the same side(s) as the chronic subdural hematoma is embolized with liquid embolic agents.
  Arms: Embolization of middle meningeal artery
Procedure: Standard neurosurgical hematoma evacuation — Standard neurosurgical evacuation of chronic subdural hematoma through burr-hole or mini craniotomy and postoperative subdural or subgaleal drainage.
  Other Names: burr-hole, mini craniotomy
  Arms: Standard neurosurgical hematoma evacuation and drainage

SUMMARY:
The SWEMMA trial is an open, national, multi-center, prospective, randomized (1:1), superiority trial designed to assess impact on reoperation rates for chronic subdural hematoma with a head-to-head comparison of embolization of the middle meningeal artery (intervention) with standard neurosurgical hematoma evacuation (control).

DETAILED DESCRIPTION:
Introduction: Chronic subdural hematoma (CSDH) is one of the most common neurosurgical disorders and the incidence is rising. The mainstay of treatment is neurosurgical hematoma evacuation followed by postoperative drainage but recurrence and reoperation rates are as high as 10-30%. Embolization of the middle meningeal artery (EMMA) has been proposed as an adjunct or as sole therapy and initial data suggests markedly reduced reoperation rates. Several randomised trials are currently underway, mostly randomizing with EMMA as an adjunctive to evacuation, or as an alternative to conservative treatment. This trial aims to make a head-to-head comparison of neurosurgical evacuation versus EMMA.

Aims: The primary objective of the trial is to compare efficacy of EMMA on rates of reoperation by randomizing patients with CSDH and mild to moderate symptoms to either EMMA or standard neurosurgical evacuation. Secondary objectives include all complication rate, technical success rate, residual hematoma volume at 3 months, neurological functionality and quality of life at 3 and 12 months and composite endpoint of death or reoperation at 3 and 12 months.

Method: Patients with previously untreated CSDH admitted to the neurosurgical unit at participating centers with clinical and/or radiological indication for neurosurgical evacuation, mild to moderate symptoms and able to provide informed consent, will be randomized to either standard treatment or EMMA. Immediately after either procedure the participant returns to standard clinical care. At 3 months a CT of the head is performed. A structured telephone interview is held by a treatment-blinded outcomes assessor at 3 months and 12 months, measuring quality of life (EQ-5D) and neurological disability (mRS). Medical records are collected and assessed at 3 months regarding safety measures. Data on reoperation and mortality are collected from the National Board of Health and Welfare and National Cause of Death Registry at 3 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18-89 y/o
2. Non-contrast Computed Tomography (NCCT)- or Magnetic Resonance Imaging (MRI)- verified, previously unoperated uni- or bilateral cSDH
3. Clinical and/or radiological status indicating neurosurgical treatment
4. Markwalder Scale score <2
5. Glasgow coma Scale score >13
6. Able to provide signed informed consent

Exclusion Criteria:

1. Acute subdural hematoma
2. Focal, non-hemispheric cSDH
3. Midline shift >10 mm and/or effaced basal cisterns and/or significant dilatation of one or both lateral ventricle temporal horns and/or incipient uncal herniation
4. Structural pathology causing the cSDH (e.g. dural AV-fistula, AVM, tumor, arachnoid cyst, ventriculoperitoneal shunt)
5. Contraindications to angiography
6. Dependency defined as mRS >3
7. Life expectancy <6 months
8. Comorbidity deemed making follow up impossible
9. Participation in other interventional clinical study
10. Pregnancy

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Reoperation | 3 months
  Reoperation rate of CSDH between groups

SECONDARY OUTCOMES:
Neurological disability | 3 months and 12 months
  Assessed by the modified Rankin Scale (mRS). Numerical scale with scores between 0 and 6 (0 = no symptoms, 6= death)
Quality of Life (EQ-5D) | 3 months and 12 months
  Assessed by the EuroQol EQ-5D scale
Residual hematoma volume | 3 months
  Change in hematoma volume from pre-, post operative, and follow up head CT
Technical success rate | 24 hours
  Rate of technically successful embolizations performed
Procedure related complication rate (Safety) | 3 months
  Difference in number and severity of complications between endovascular and surgical participants
Composite endpoint | 3 and 12 months
  Death or reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Drake, MD, Principal Investigator — Skåne University Hospital, Lund University, Lund Sweden; Johan Wassélius, MD, PhD, Study Director — Skåne University Hospital, Lund University, Lund Sweden
Locations (4):
- Sweden (4):
  - Sahlgenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Karolinska Hospital, Stockholm
  - Norrlands Universitetssjukhus, Umeå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drake M, Ullberg T, Nittby H, Marklund N, Wasselius J. Swedish trial on embolization of middle meningeal artery versus surgical evacuation in chronic subdural hematoma (SWEMMA)-a national 12-month multi-center randomized controlled superiority trial with parallel group assignment, open treatment allocation and blinded clinical outcome assessment. Trials. 2022 Nov 8;23(1):926. doi: 10.1186/s13063-022-06842-4. PMID 36348417